CLINICAL TRIAL: NCT00837122
Title: Genetics of Type 2 Diabetes in Diverse Populations
Brief Title: Genetics of Type 2 Diabetes in West Africans
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909070; 09-HG-N070
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-09-05

CONDITIONS: Hypertension; Diabetes
Keywords: African; Natural History
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Control subjects are nondiabetics ethnically matched to patients
- T2D: Patients with confirmed T2D who are newly diagnosed or on treatment in Ibadan, Nigeria

SUMMARY:
Background:

* Type 2 diabetes (T2D) and associated complications are major contributors to the global disease burden. T2D is already a major health threat in populations in developed countries and is rapidly taking hold in the developing world.
* It is believed that understanding the complex interplay between genetic and lifestyle characteristics in the etiology of T2D and related complications will lead to the development of better preventive and therapeutic strategies. In Addition, the results of this project will facilitate our understanding of causes of diabetes in African Americans, other US and world populations

Objectives:

* To conduct a genome-wide association study (GWAS) to identify susceptibility genetic variants for diabetes among the Yoruba people in Ibadan, Nigeria.
* To enroll and examine 300 unrelated cases of T2D and 300 ethnicity-matched Yoruba controls.
* To conduct resequencing of positional candidate gene/loci to identify likely functional variants in a subset of the cohort.
* To conduct replication studies of the top-100 scoring variants in three independent African and European ancestry samples.
* To investigate whether diabetes-associated variants discovered in European populations increase diabetes risk in West Africans.

Eligibility:

* Patients 18 years of age with confirmed T2D who are newly diagnosed or on treatment of Yoruba ethnicity in Ibadan, Nigeria. Control subjects are nondiabetics ethnically matched to patients.

Design:

* The study design for both patients and controls consists of the following steps:
* Discuss informed consent process and obtain signed informed consent form. Informed consent will be administered by trained clinic staff.
* Assign study ID (barcode)
* Administer questionnaires
* Obtain spot urine sample
* Measure blood pressure
* Obtain anthropometric measurements including body composition
* Perform finger prick for blood glucose level
* Obtain venous blood samples
* Perform eye examination
* On the following day, perform confirmatory blood glucose for the small subset of participants requiring confirmation of previous test result DNA extraction of stored samples will be done at either the National Institutes of Health or the laboratory in Nigeria.
* GWAS will be conducted using publicly available software packages.

DETAILED DESCRIPTION:
Study Description:

This protocol is designed to study the genetic basis of Type 2 Diabetes (T2D) and related conditions in Africa.

Objectives:

Primary Objective: To conduct genetic association studies of T2D, T2D complications, and related traits in Africans of diverse ethnic groups

Secondary Objectives:

* To investigate the contribution of gene x environment interactions in T2D risk and in influencing related traits
* To develop a large-scale genetic epidemiological resource for the replication of findings in other studies of related traits
* To conduct trans-ethnic fine-mapping
* To describe the study population epidemiologically in terms of cardiometabolic traits and prevalence of related conditions
* To conduct population genetic analyses to describe population history and to develop statistical techniques appropriate for genetic analyses of African ancestry individuals
* To conduct deep phenotyping to facilitate additional research questions related to cardiometabolic traits and for follow-up previous findings

Endpoints:

Primary Endpoint: T2D

Secondary Endpoints: T2D Complications, Hypertension, Obesity, Dyslipidemia, Metabolic Syndrome, Chronic Kidney Disease, and other cardiometabolic traits

ELIGIBILITY:
* INCLUSION CRITERIA:

As our primary interest is in T2D, it is important to exclude individuals who may have diabetes of another etiology. Elevated blood glucose in individuals 25 years old or younger is unlikely (in West Africa) to result from T2D and may reflect Type 1 Diabetes. Therefore, only individuals older than 25 years will be included in this study.

We are seeking to enroll persons without T2D or with previously or newly diagnosed T2D. Previously diagnosed cases will be determined by self-report of being treated with oral medication or insulin. Newly diagnosed cases will be determined by fasting blood glucose value >= 126 mg/dl on more than one occasion. Individuals who have elevated blood glucose during their initial reading will be asked to return to the study site for a second test. If this test also has a fasting blood glucose value >= 126 mg/dl, then they will be considered a new case. The control group will be individuals with no report of T2D diagnosis and fasting plasma glucose (FPG)< 126 mg/dl.

Only unrelated individuals will be included in this phase of the study to avoid confounding genetic association studies by relatedness in the study population.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Incarceration.
* Lack capacity to consent to research participation.
* Pregnancy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed T2D who are newly diagnosed or on treatment and those without T2D (ethnically matched) in Ibadan, Nigeria
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-02-03 (Actual)

PRIMARY OUTCOMES:
I | ongoing
  In a subset of participants, to investigate the relationship between diets, gut microbiota, and T2D/related traits.
H | ongoing
  To investigate whether hemoglobin A1c (HbA1c) as an indicator of blood glucose control over time is reliable in the presence of the sickle cell trait (HbS), a common hemoglobinopathy in West Africa. The association between HbA1c repeated measures and changes in T2D-related traits over time will be evaluated. We will also evaluate if there is a systematic difference (bias) in the estimation of A1c in carriers of the sickle trait and non-carriers in persons with and without diabetes.
G | ongoing
  g- In a subset of participants, to investigate key tissues in the pathophysiology of T2D, we will study differences in the gene expression of skeletal muscle and adipose tissue in lean and obese individuals with and without T2D (n=100, Biopsy Substudy).
F | ongoing
  f- To conduct population genetic analyses to describe population history and to develop statistical techniques appropriate for genetic analysis of African ancestry individuals.
E | ongoing
  e-To describe these individuals epidemiologically in terms of metabolic traits and the prevalence of relevant conditions, as, for some traits, this may be the first large-scale epidemiological, population-based study of Africans with the appropriate data for such description.
D | ongoing
  d- To conduct trans-ethnic fine mapping to determine whether the reduced LD across the genome in African ancestry individuals can refine the region of interest around genetic associations discovered in populations of non-African ancestry. To conduct candidate gene resequencing, Whole Genome Sequencing (WGS), or Whole Exome Sequencing (WES), as funding allows, in participants with metabolic profiles of interest. For instance, individuals will be selected who have extreme values for serum lipids for WES. Variants identified by this resequencing will be genotyped in the larger study population for association analysis.
C | ongoing
  c- To develop a large-scale genetic epidemiological resource for the replication of findings in other studies of related traits in African ancestry and non-African ancestry individuals.
B | ongoing
  b- To investigate the contribution of gene x environment interactions in T2D risk and in influencing related traits. These investigations may be conducted on either a hypothesis-driven, locus-specific manner or agnostically, i.e. genome-wide. Environmental variants to be considered include lifestyle factors (e.g. diet, measured by food frequency questionnaires (FFQ), socioeconomic measures, and medications taken.
A | ongoing
  a- To conduct genetic association studies of T2D and related traits (including blood pressure, serum lipids, blood glucose, adiposity) in West Africans of diverse ethnic groups. Approaches will include genome-wide association studies (including exome chip data) and candidate gene/loci association analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Rotimi, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (5):
- Ghana (2):
  - University of Ghana, Accra
  - University of Science and Tech, Kumasi
- Nigeria (3):
  - University of Nigeria, Enugu
  - University of Ibadan, Ibadan
  - University of Lagos, Lagos

IPD SHARING:
Plan to Share IPD: No
Extensive review of the consents related to this protocol by the NHGRI IRB was conducted and it was determined that because the initial consent process did not address sharing of participants' data and the related risks and the carefully established rapport and trust with African populations and collaborators, it would not be appropriate to share participant's data. A memorandum to this effect can be provided, if necessary. We will continue to be open to making the data available through collaboration, a use of the data that was described in initial consent forms.